CLINICAL TRIAL: NCT07368842
Title: Scalp Hair Metabolomics as a Novel Biomarker of Poor Metabolic Health in Individuals With Severe Obesity
Brief Title: Scalp Hair Metabolomics in Severe Obesity
Status: Not yet recruiting | Type: Observational
Sponsor: Singapore General Hospital (Other)
Responsible Party: Principal Investigator, Tan Hong Chang, Dr, Singapore General Hospital
Other Study IDs: SGH_Hair01_2025
Record Dates: First submitted 2026-01-20; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Obesity & Overweight; Hair Loss; Metabolomics; Bariatric Surgery
Keywords: obesity; hair loss; metabolomics; bariatric surgery
MeSH Terms: conditions — Obesity; Overweight; Alopecia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — hair samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy control: Healthy control with normal weight
- Severe obestiy: Severe obesity

SUMMARY:
The purpose of this research study is to investigate how body weight and weight-loss surgery affect the natural chemicals found in scalp hair over time. We will also find out how common and severe hair thinning/hair loss and muscle loss are in the first 6 months after bariatric surgery.

DETAILED DESCRIPTION:
We will recruit 30 subjects with severe obesity scheduled for bariatric surgery and 30 healthy-weight controls.

Following written informed consent, we will collect the study subject's medical information, conduct a dietary and quality-of-life survey, take body measurements, obtain scalp photos, perform a hair-pull test, collect a hair sample, and conduct muscle strength testing. Controls will be assessed only at baseline. Those with severe obesity will return at 4 ± 2 weeks, 12 ± 4 weeks, and 26 ± 4 weeks following bariatric surgery to repeat the study procedures.

ELIGIBILITY:
Inclusion Criteria:

All subjects:

1. Age 21-70 years
2. Ability to provide informed consent

Healthy weight controls:

1. BMI of 18.5-24.9 kg/m2
2. No chronic disease
3. No long-term medications

Severe obesity:

1. BMI of > 32.5 kg/m2
2. Scheduled to undergo bariatric surgery

Exclusion Criteria:

1. Pregnancy
2. Any factors likely to limit adherence to study protocol
3. Any history of autoimmune or scarring alopecia (eg. alopecia areata, discoid lupus, lichen planopilaris)

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with severe obesity will be recruited from the Singapore General Hospital's obesity clinic, while controls will be healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2026-02-07 (Estimated); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Amino acid concentration | From enrollment to the end of study duration at 6 months
  Post-surgery changes in scalp hair amino acid concentration following bariatric surgery

SECONDARY OUTCOMES:
Severity of hair loss | From the time of enrolment until the end of the study at 6 months
  The severity of hair loss is measured by quantifying the number of hairs lost during the hair pull test
Scalp hair amino acid concentration (between groups) | At the time of enrollment
  Differences in scalp hair amino acid concentration between controls and those with severe obesity
Grip strength | From enrollment until the end of the study at 6 months
  The post-surgery changes in grip strength measured using handgrip dynamometer
Sit to stand speed | From enrollment until study completion at 6 months
  Time taken to complete sit to stand test after bariatric surgery
Hair specific Skindex-29 score | From enrollment until study completion at 6 months
  Hair specific Skindex-29 quality of life questionnaire score after bariatric surgery

CONTACTS AND LOCATIONS:
Overall Officials: Hong Chang Tan, Principal Investigator — Singapore General Hospital

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication